CLINICAL TRIAL: NCT02852460
Title: The Influence of Rapid Recovery on Sleep Quality Following Total Hip Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Yang, Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Rapid recovery
Record Dates: First submitted 2016-07-24; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Arthroplasty; Recovery of Function; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

ARMS (2):
- Experimental group (Experimental): rapid recovery
  Interventions: Other: rapid recovery
- Controlled group (No Intervention): non-rapid recovery

INTERVENTIONS:
Other: rapid recovery
  Arms: Experimental group

SUMMARY:
To evaluate the influence of rapid recovery on sleep quality following total hip replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary unilateral total hip arthroplasty;
* 2. Patients with hip osteoarthritis,rheumatoid arthritis or femoral head necrosis;
* 3. Able and willing to provide signed informed consent.

Exclusion Criteria:

* 1. Simultaneously bilateral total hip arthroplasty or revision case;
* 2. Surgical History of the hip joint;
* 3. Hip joint cavity paracentesis in recent 3 months;
* 4. Stiffness with hip;
* 5. Blood coagulation disorders;
* 6. History of deep venous thrombosis;
* 7. Concomitant medical problems such as uncontrolled hypertension, severe cardiovascular disorder, chronic obstructive pulmonary disease, liver or renal failure
* 8. Allergic to NSAIDs, opioid analgesics, zolpidem
* 9. Sleep apnea, Parkinson disease, dementia, depression
* 10. Use of sedatives or hypnotics
* 11. Unable to comply with polysomnographic measurement

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the pain, stiffness and joint function of operated limb by McMaster Universities Osteoarthritis Index(WOMAC) | 6 months
  To evaluate the function and structure of hip joint from the aspect of pain, stiffness and joint function
To evaluate the anxiety of patients post-operation by Generalized Anxiety Disorder scale-7 (GAD-7) | 6 months
To evaluate the sleep quality of patients post-operation by Pittsburgh Sleep Quality Index (PSQI) | 6 months
Insomnia severity index | 6 months
To evaluate the health related quality of life of patients post-operation by the 12-items Short Form Health Survey (SF-12) | 6 months
To evaluate the pain severity of patients post-operation by Visual Analogue Scale (VAS) Pain Score | 6 months

SECONDARY OUTCOMES:
C Reactive Protein (CRP) | 6 months
Erythrocyte Sedimentation Rate (ESR) | 6 months
To evaluate the quadriceps strength according to grade division standard published by British Medical Research Council | 6 months
To evaluate the swelling of operated limb by measure the thigh girth increment | 6 months
  Calculated by operated limb thigh girth increment post-operation
To evaluate the operation satisfaction of patients by Visual Analogue Scale (VAS) Satisfaction Score | 6 months
To evaluate the function of operated limb by Harris hip score (HHS) | 6 months
To evaluate the range of motion (ROM) of operated hip | 6 months
  ROM of operated hips post-operation
Length of hospital stay | 3 months
Number of dressing changes | 1 month
  Number of dressing changes post-operation
Hematocrit | 6 months
  Pre-operation and post-operation hematocrit
Haemoglobin | 6 months
  Pre-operation and post-operation haemoglobin
Number of Blood transfusion cases | 1 month
Blood transfusion volume | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China